CLINICAL TRIAL: NCT01820559
Title: Efficacy and Safety of Eslicarbazepine Acetate as Preventive Therapy for Subjects With Migraine: a Doubleblind,Randomised, Placebo-controlled, Parallel-group, Multicentre Clinical Trial
Brief Title: Efficacy and Safety of Eslicarbazepine Acetate as Preventive Therapy for Subjects With Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-2093-209
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-04

CONDITIONS: Migraine
Keywords: migraine; ESL; eslicarbazepine acetate
MeSH Terms: conditions — Migraine Disorders | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ESL 1200 mg (Active Comparator): eslicarbazepine acetate 1200 mg
  Interventions: Drug: ESL 1200 mg
- ESL 800 mg (Active Comparator): eslicarbazepine acetate 800 mg
  Interventions: Drug: ESL 800 mg
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Tablets
  Other Names: Sugar pills
  Arms: Placebo
Drug: ESL 1200 mg — Eslicarbazepine acetate was supplied in 400-mg and 600-mg tablets and was administered with a dose of 800 or 1200 mg QD in the evening by the oral route.
  Other Names: Eslicarbazepine acetate
  Arms: ESL 1200 mg
Drug: ESL 800 mg — Eslicarbazepine acetate was supplied in 400-mg and 600-mg tablets and was administered with a dose of 800 or 1200 mg QD in the evening by the oral route.
  Other Names: Eslicarbazepine acetate
  Arms: ESL 800 mg

SUMMARY:
This was a multinational, randomised, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy, safety, and tolerability of multiple doses of ESL as prophylactic treatment in subjects with migraine with or without aura. Subjects were randomised in a 1:1:1 ratio to receive placebo, ESL 800 mg/day once daily (QD), or ESL 1200 mg/day QD.

DETAILED DESCRIPTION:
The study consisted of a Screening Period of 2 to 4 weeks, a 4-week placebo Baseline Period, a 2-week Titration Period, a 12-week Maintenance Period, and a 4-week Follow-up Period. During the entire study the subjects had a diary to document the occurrence, duration, and intensity of headaches, the occurrence or not of aura and its nature, as well as other related symptoms, and the use of study medication and acute medication.

ELIGIBILITY:
Inclusion Criteria:

* Women or men, 18 years of age or older (according to Amendment #1 for Czech Republic [24 Mar 2009]: 18 to 65 years of age).
* Diagnosis (established prior to 50 years of age) of migraine headaches for at least 1 year, and a well-documented history of migraine headaches with or without aura according to the criteria of the IHS (see Section 3.5.6.1) for at least 3 months (according to Amendment #1 for Czech Republic [24 Mar 2009]: for at least 3 months with at least 3 migraine attacks per month in each of these 3 months).
* At least 2 (according to Amendment #1 for Czech Republic [24 Mar 2009]: at least 3) (and no more than 10) well-defined migraine headache attacks per month, with at least 24 h of freedom from headaches and other symptoms of migraine between attacks.
* Able to distinguish the migraine headache attacks from other types of common headaches (tension-type headaches, sinus-related headaches, etc.).
* Not taking any prophylactic migraine therapies for at least 2 weeks prior to Baseline Visit (V2). Flunarizine had to be discontinued at least 4 weeks prior to V2.
* Able and willing to provide written informed consent to participate in the study after having the opportunity to review the Subject Information Sheet and Informed Consent Form (ICF).
* Able and willing to comply with all study requirements, in the judgment of the investigator.
* Women were surgically sterile (i.e. bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or at least 2 years postmenopausal or, if of childbearing potential, were sexually abstinent or agreed to use medically acceptable non-hormonal methods of contraception (see Section 3.3.3). (According to Amendment #1 for Czech Republic [24 Mar 2009]: Women were sexually abstinent or agreed to use a double-barrier method of contraception. Hormonal contraceptives were not acceptable as a contraceptive method in this study. However, their intake was not forbidden throughout the study.)

Exclusion Criteria:

* A known hypersensitivity to ESL or to other carboxamide derivatives (e.g. oxcarbazepine, carbamazepine), or to any of the excipients.
* Suspected or confirmed medication-overuse headache.
* More than 14 headache days (migraine or other headache types) per month in either of the 2 months prior to screening.
* Consistent or recurrent frequent headaches (i.e. ≥6 headache days a month) other than migraine headaches.
* Unable to discontinue medications primarily used for migraine prophylaxis that have been commonly used for other indications (tricyclic agents, divalproic acid, topiramate, etc.). A subject who received beta blockers or calcium channel blocker therapy for reasons other than migraine prophylaxis was eligible for inclusion, provided his/her dosing regimen had been stable for ≥2 months and was not expected to change during the course of the study.
* Using prohibited concomitant medication (see Section 3.5.5.2).
* A white blood cell (WBC) count <2.5 * 109/L, neutrophil count <1.5 * 109/L, sodium <125 mmol/L, or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥2 times the upper limit of normal at V1 (Screening Visit), or any other clinically relevant laboratory abnormality that, in the investigator's opinion, could compromise the subject's safety.
* A creatinine clearance lower than 60 mL/min at screening.
* A second- or third-degree atrioventricular blockade not corrected with a pacemaker or any other clinically significant abnormality in the 12-lead electrocardiogram (ECG) as determined by the investigator.
* Pregnant or nursing women.
* A history of chronic alcohol or drug abuse or addiction within the last 2 years.
* A severe hepatic, renal, respiratory, haematological, or immunologic illness, unstable cardiovascular disease, or any other medical or psychiatric condition that, in the judgment of the investigator, made the subject inappropriate for entry into this study.
* Received an investigational drug (or a medical device) within 3 months of screening or was currently participating in another study of an investigational drug (or medical device).
* An employee of the investigator or study centre, with direct involvement in the proposed study or other studies under the direction of that investigator or study centre, or was a family member of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Soares-da-Silva, MD, PhD, Study Director — BIAL - Portela & Ca. SA

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablets
  Placebo : Tablets
- ESL 800 mg: eslicarbazepine acetate 800 mg
  ESL 800 mg :
- ESL 1200 mg: eslicarbazepine acetate 1200 mg
  ESL 1200 mg :
Period: Overall Study
Arm/Group | Placebo | ESL 800 mg | ESL 1200 mg
Started | 136 | 135 | 139
Randomized and Treated | 136 | 135 | 139
Completed Tutration Period | 130 | 134 | 131
Entered Maintenance Period | 129 | 133 | 129
Completed Maintenance Period | 122 | 123 | 110
Completed | 122 | 122 | 110
Not Completed | 14 | 13 | 29
Not completed — Adverse Event | 4 | 6 | 13
Not completed — Withdrawal by Subject | 1 | 2 | 5
Not completed — Protocol Violation | 2 | 1 | 3
Not completed — Subject's non-compliance | 1 | 0 | 2
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — At sponsor request | 0 | 0 | 1
Not completed — Lack of Efficacy | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ESL 800 mg | ESL 1200 mg | Total
Number analyzed (Participants) | 136 | 135 | 139 | 410
Age, Customized [Number; unit: participants]
  <=65 years | 135 | 135 | 136 | 406
  >65 years | 1 | 0 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 114 | 111 | 346
  Male | 15 | 21 | 28 | 64

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in the Frequency of Migraine Attacks
Description: The primary efficacy variable was the absolute change from baseline in the frequency of migraine attacks standardised to 4 weeks in the Maintenance Period, as recorded in the subject diary. If there were less than 24 h between the end of 1 migraine event and the start of the next event, these 2 events were considered to belong to 1 migraine attack. There had to be a minimum of 24 h of freedom from headache, pain, and symptoms of migraine between attacks recorded in the subject diary to be considered as more than 1 attack of migraine for statistical analysis.
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: number of migraine attacks/participant
Arm/Group | Placebo | ESL 800 mg | ESL 1200 mg
Number analyzed (Participants) | 133 | 134 | 136
number of migraine attacks/participant | -0.8 (0.1429) | -1.0 (0.1428) | -1.0 (0.1416)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events(TEAEs) were evaluated throughout the study TEAEs, i.e. those Adverse Events (AEs) starting after the first dose intake until 28 days after the last dose, have been summarised by SOC and PT
Arm/Group | Placebo | ESL 800 mg | ESL 1200 mg
Serious Adverse Events (participants affected / at risk) | 1/136 | 1/135 | 4/139
Other Adverse Events (participants affected / at risk) | 46/136 | 67/135 | 74/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=136) | ESL 800 mg (N=135) | ESL 1200 mg (N=139)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
STATUS MIGRAINOSUS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=136) | ESL 800 mg (N=135) | ESL 1200 mg (N=139)
Dizziness (Nervous system disorders) | 2 (2) | 6 (6) | 14 (14)
Somnolence (Nervous system disorders) | 1 (1) | 9 (9) | 13 (13)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 4 (4) | 11 (11)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (6) | 10 (10)
Migraine (Nervous system disorders) | 3 (3) | 2 (2) | 6 (6)
Nasopharyngitis (Infections and infestations) | 6 (6) | 5 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3)
Fatigue (General disorders) | 1 (1) | 4 (4) | 3 (3)
Influenza (General disorders) | 2 (2) | 3 (3) | 3 (3)
Asthenia (General disorders) | 0 (0) | 2 (2) | 3 (3)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Status migrainosus (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
Face oedema (General disorders) | 0 (0) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 2 (2) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 1 (1)
Insomnia (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other